CLINICAL TRIAL: NCT06800196
Title: A Phase I, Multicenter, Open-label Study to Evaluate the Safety, Pharmacokinetics, Preliminary Efficacy of KNT-0916 in Subjects with Unresectable or Metastatic Solid Tumors with FGFR2 Alterations
Brief Title: A Study of KNT-0916 in Treatment of Unresectable or Metastatic Solid Tumors with FGFR2 Alterations
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: KinoTeck Therapeutics Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EO002-CP002
Record Dates: First submitted 2025-01-20; First posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Solid Tumors with FGFR2 Alterations, Adult

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part A - dose escalation (Experimental): Dose escalation of KNT-0916 in patients with advanced solid tumors.
  Interventions: Drug: KNT-0916
- Part B - expansion (Experimental): Oral dose of KNT-0916 as determined during Part A Dose Escalation.
  Interventions: Drug: KNT-0916

INTERVENTIONS:
Drug: KNT-0916 — • KNT-0916 is an oral inhibitor of FGFR2.

SUMMARY:
This is a Phase1, open-label, dose escalation and expansion study designed to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics and preliminary efficacy of KNT-0916 in patients with unresectable or metastatic solid tumors harboring FGFR2 alterations who have failed prior systemic therapy. This study is divided into 2 parts, dose escalation part(part A), dose expansion part(partB).

DETAILED DESCRIPTION:
This study is divided into 2 parts, part a isNdesigned to explore the maximum toxicity dose (MTD) of KNT-0916 with an accelerated titration plus traditional "3+3" design; part b is designed to explore the elementary anti-neoplastic activity of KNT-0916 with recommended dose in patients with confirmed FGFR2 alterations through central laboratory testing.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed unresectable or metastatic solid tumor
* Documented FGFR2 gene fusion, mutation, or amplification per testing of blood and/or tumor
* Patient must have measurable disease per RECIST v1.1
* Patient has ECOG performance status of 0-1
* Patient must have disease that is refractory to standard therapy, disease that has not adequately responded to standard therapy, disease for which standard or curative therapy does not exist, or the patient must be intolerant to or have declined standard therapy
* An expected survival of ≥ 12 weeks.
* Adequate organ function, as measured by laboratory values

Exclusion Criteria:

* Prior treatment with any FGFR2 target therapy.
* Central nervous system metastasis with associated symptom and signs.
* Clinically significant, uncontrolled cardiovascular disease.
* History of interstitial lung disease, or infectious pneumonitis need heavy antibiotics therapy 5. As judged by the investigator, unsuitable for attending the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Estimated)
Dates: Start 2025-03-31 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting Toxicity (DLT) | 4 weeks
Maximum tolerated dose (MTD) or Maximum administered dose (MAD) | 12 months
Incidence, relatedness, seriousness and severity of adverse events (AEs) per the National Cancer Institute Common Terminology Criteria for AE (NCI CTCAE) Version 5.0. | 33 months
Recommended phase 2 dose (RP2D) | 33 months

SECONDARY OUTCOMES:
Objective response rate (ORR) assessed as per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 | 33 months
Duration of response (DoR) assessed as per RECIST 1.1 | 33 months
Disease control rate (DCR) assessed as per RECIST 1.1 | 33 months
Progression-free survival (PFS) assessed as per RECIST 1.1 | 33 months
Overall survival (OS) assessed as per RECIST 1.1 | 33 months
Pharmacokinetic parameters including maximum plasma drug concentration (Cmax) | 33 months
Pharmacokinetic parameters including area under the plasma concentration versus time curve (AUC) | 33 months
Pharmacokinetic parameters including half-life (t1/2) | 33 months
Pharmacokinetic parameters including time to maximum concentration (Tmax) | 33 months
Pharmacokinetic parameters including Apparent clearance (CL/F) | 33 months

CONTACTS AND LOCATIONS:
Overall Officials: Ruihua Xu, Principal Investigator — Sun Yat-sen University

IPD SHARING:
Plan to Share IPD: No